CLINICAL TRIAL: NCT04359836
Title: A Non-Interventional Pilot Study to Explore the Role of Gut Flora in COVID-19 Infection
Brief Title: A Study to Explore the Role of Gut Flora in COVID-19 Infection
Status: Recruiting | Type: Observational
Sponsor: ProgenaBiome (Other)
Responsible Party: Sponsor
Other Study IDs: PRG-041
Record Dates: First submitted 2020-04-20; First posted 2020-04-24 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Gut Microbiome; Gastrointestinal Microbiome; COVID; COVID-19; Corona Virus Infection; Coronavirus; Coronaviridae Infections; Coronavirus 19; Coronavirus-19; COVID 19
Keywords: Microbiome; Coronavirus; Corona Virus; 19; COVID; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections; Coronaviridae Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Stool samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- General Population: The general population will have their microbiome sequenced from stool samples provided.
  Interventions: Other: There is no intervention in this study

INTERVENTIONS:
Other: There is no intervention in this study — There is no intervention in this study

SUMMARY:
This study seeks to determine whether the virus which causes COVID-19, SARS-CoV-2, is shed in the stools of patients who are infected.

DETAILED DESCRIPTION:
In this study the stool of patients who are being treated for COVID-19 will be tested during treatment and then again following treatment to determine if the virus is shed in the stool during infection, afterwards, or both.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, demonstrating that the patient understands the procedures required for the study and the purpose of the study
2. Male or female of 18 years of age or older
3. Diagnosis of COVID-19 infection by RT- PCR within 1 week of Screening

Exclusion Criteria:

1. Refusal to sign informed consent form
2. History of bariatric surgery, total colectomy with ileorectal anastomosis or proctocolectomy.
3. Postoperative stoma, ostomy, or ileoanal pouch
4. Treatment with total parenteral nutrition

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults 18 and older
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-04-16 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Correlation of Microbiome to Disease via Relative Abundance Found in Microbiome Sequencing | One year
  Relative abundance of bacterial classes within taxonomic phyla and, more broadly, within their domain will be analyzed by sequencing the gut microbiome. These data will then be categorized among specific gastrointestinal disease types.

SECONDARY OUTCOMES:
Validation of Sequencing Methods | One year
  To validate the methods used to sequence samples

CONTACTS AND LOCATIONS:
Overall Officials: Sabine Hazan, MD, Principal Investigator — ProgenaBiome
Locations (1):
- ProgenaBiome, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papoutsis A, Borody T, Dolai S, Daniels J, Steinberg S, Barrows B, Hazan S. Detection of SARS-CoV-2 from patient fecal samples by whole genome sequencing. Gut Pathog. 2021 Jan 30;13(1):7. doi: 10.1186/s13099-021-00398-5. PMID 33516247